CLINICAL TRIAL: NCT00567827
Title: Identification of Bacterial Species and Their Antibiotic-Resistant Spectrum in Sputum Specimen From the Patients With Pneumonia Via Nuclear Acid Detection Assay
Brief Title: Pathogen Identification of Bacterial Pneumonia Via DNA Detection
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Professor Zhancheng Gao,, Peking University People's Hospital
Other Study IDs: 2006AA02Z4A9; 2006AA02Z4A9 (Other Grant/Funding Number: the National Hi-Tech Project of P.R. China)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Pneumonia
Keywords: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from sputum specimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pneumonia is a common cause of morbidity and mortality. The diagnosis of pneumonia from the microbiology perspective has been challenging. Recent reports suggest the utility of nuclear acid detection for rapid and accurate diagnoses of these pathogens and their antibiotic-resistant spectrum. Extracted bacterial nucleic acid in sputum specimen will be identified by Nuclear acid detection assay kit with Microfluidic Pumping Chip and LAMP methods

DETAILED DESCRIPTION:
Sputum specimens normally collected from the patients with pneumonia for routine microbiologic testing and extra specimens will be evaluated via nuclear acid assay developed in our laboratory. The assay will be directed at variety of both pathogens, including Streptococcus pneumoniae, Hemophilus influenzae, Klebsiella pneumoniae, Staphylococcus aureus, Pseudomonas aeruginosa, Acinetobacter, Mycoplasma pneumonia, Chlamydia pneumoniae and Legionella pneumophila, and common antibiotic-resistant genes, such as ESBLs genes, MecA, OprD. The ultimate goal is to have an available panel of highly accurate and rapid (same day) assay, which will be carried out in several hours for identification.

The extracted pathogen nucleic acid in sputum specimen will be identified by Nuclear acid detection assay with Microfluidic Pumping Chip and LAMP methods. The species of bacteria and their antibiotic-resistant gene to be detected are as listed above. As nucleic acid extracts will be archived, other pathogens can be investigated in the future if the correlated assay is developed. All results obtained by nuclear acid detection will be compared to results for conventional testing as listed above. Sensitivity, specificity and predictive values will be calculated. In cases where discordant results occur, additional testing and or medical history review will be properly conducted.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age.
* Cough present greater than one day
* History of fever
* X-ray evidence of pneumonia.

Exclusion Criteria:

* Pneumonia caused by TB, fungi and virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greater than 18 years of age. Cough present greater than one day and a history of fever and X-ray evidence of pneumonia.
Sampling Method: Probability Sample
Enrollment: 2896 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhancheng Gao, Professor, Principal Investigator — Peking University People's Hospital

REFERENCES:
- [Derived] Kang Y, Deng R, Wang C, Deng T, Peng P, Cheng X, Wang G, Qian M, Gao H, Han B, Chen Y, Hu Y, Geng R, Hu C, Zhang W, Yang J, Wan H, Yu Q, Wei L, Li J, Tian G, Wang Q, Hu K, Wang S, Wang R, Du J, He B, Ma J, Zhong X, Mu L, Cai S, Zhu X, Xing W, Yu J, Deng M, Gao Z. Etiologic diagnosis of lower respiratory tract bacterial infections using sputum samples and quantitative loop-mediated isothermal amplification. PLoS One. 2012;7(6):e38743. doi: 10.1371/journal.pone.0038743. Epub 2012 Jun 14. PMID 22719933